CLINICAL TRIAL: NCT00004084
Title: Phase I/II Radioimmunotherapy of Non-Hodgkin's Lymphoma With Radiolabeled Humanized Immu-LL2: Treatment With 90Y-hLL2 IgG
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Lymphoma or Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Garden State Cancer Center at the Center for Molecular Medicine and Immunology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert M Sharkey, GSCC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067295; R01CA067026 (NIH); CMMI-C-037A-97; NCI-H99-0041; NCI-V99-1567
Record Dates: First submitted 1999-12-10; First posted 2004-04-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Leukemia; Lymphoma
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Indium

INTERVENTIONS:
Radiation: indium In 111 LL2 IgG — single dose, intravenous infusion over 30 minutes
Radiation: yttrium Y 90 epratuzumab — single dose, intravenous infusion over 30 minutes

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate cancer cells and deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody therapy in treating patients who have lymphoma or leukemia that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and dose limiting toxicity of yttrium Y 90-labeled humanized anti-CD22 monoclonal antibody LL2(90Y-hLL2 IgG) in patients with B-cell malignancies. II. Determine the pharmacokinetics and biodistribution of indium In 111 humanized LL2 (111In-hLL2 IgG) in these patients. III. Evaluate the immunogenicity of repeated injections of 90Y-hLL2 IgG in these patients. IV. Determine whether 90Y-hLL2 IgG versus indium In 131 humanized LL2 IgG has a therapeutic advantage based on organ and tumor dosimetry obtained with 111In-hLL2 IgG.

OUTLINE: This is a dose escalation study. Patients are stratified into risk groups (high vs low). Patients receive pretherapy imaging with indium In 111 humanized LL2 IgG IV for up to 30 minutes on days -7 to 0. Patients receive yttrium Y 90-labeled humanized anti-CD22 monoclonal antibody LL2 (90Y-hLL2-IgG) IV for up to 30 minutes on day 0. Cohorts of 3-6 patients receive escalating doses of 90Y-hLL2-IgG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding the dose at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. Patients are followed every 2 weeks for 1 month, monthly for 2 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed B-cell malignancy, including B-cell non-Hodgkin's lymphoma or B-cell chronic lymphocytic leukemia, that has failed at least one regimen of standard chemotherapy At least 1 confirmed tumor site by radiolabeled LL2 IgG No greater than 25% bone or bone marrow involvement No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL AST and alkaline phosphatase less than 1.5 times upper limit of normal (ULN) (except for bone involvement) Renal: Creatinine less than 1.5 times ULN Other: Not pregnant Fertile patients must use effective contraception during and for 3-6 months after study HIV negative No severe anorexia, nausea, or vomiting No other significant concurrent medical condition that would interfere with compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior murine monoclonal antibody therapy allowed (if unreactive to yttrium Y 90-labeled humanized anti-CD22 monoclonal antibody LL2 by HPLC or ELISA test) Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: At least 2 weeks since prior corticosteroids (except for adrenal insufficiency) Radiotherapy: At least 4 weeks since prior radiotherapy to the index lesion No prior extensive radiotherapy to greater than 25% of bone marrow (except total body irradiation as part of bone marrow or stem cell transplantation regimen with engraftment of functional marrow (i.e., producing normal peripheral blood counts) No prior maximum tolerated dose levels of radiotherapy to critical organs (e.g., lung, liver, or kidney) Surgery: At least 4 weeks since prior major surgery Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 1998-04; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Burton, MD, Study Chair — Garden State Cancer Center at the Center for Molecular Medicine and Immunology
Locations (2):
- United States (2):
  - Garden State Cancer Center, Belleville, New Jersey
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania